CLINICAL TRIAL: NCT03977116
Title: Clinical Outcomes and Long Term Effects of Sodium-glucose Co-transporter 2 Inhibitors in Diabetes Mellitus and Failing Heart Patients With Implantable Cardioverter Defibrillator Undergoing Trans-catheter Ablation for Ventricular Arrhythmias.
Brief Title: Sodium-glucose Co-transporter 2 Inhibitors Effects in Failing Heart Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, clinical professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SecondUNI 05.06.2019
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus; Heart Failure; Ventricular Arrythmia
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- heart failure patients with diabetes treated by SGLT2 drugs (Experimental): Patients affected by heart failure and diabetes mellitus. These patients previous received an internal cardioverter defibrillator (ICD), and then a catheter ablation for ventricular arrhythmias (VA) therapy. After CA these patients received SLGT2 therapy.
  Interventions: Drug: SLGT2
- heart failure patients with diabetes treated by placebo (Placebo Comparator): Patients affected by heart failure and diabetes mellitus. These patients previous received an internal cardioverter defibrillator (ICD), and then a catheter ablation for ventricular arrhythmias (VA) therapy. After CA these patients received placebo therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLGT2 — These patients will receive SLGT2 therapy after catheter ablation.
  Arms: heart failure patients with diabetes treated by SGLT2 drugs
Drug: Placebo — These patients will receive placebo therapy after catheter ablation.
  Arms: heart failure patients with diabetes treated by placebo

SUMMARY:
SLGT2 therapy is safety used in heart failure (HF) patients with depressed left ventricle ejection fraction (LVEF) and diabetes mellitus (DM). These patients experience higher rate of ventricular arrhythmias (VA), that are a leading cause of cardiac arrest and mortality. However, these patients are treated by implantable cardioverter defibrillator (ICD) and cardiac resynchronization with defbrillator devices (CRTd) implant. In this setting, the catheter ablation (CA) treatment has been used to reduce the ventricular arrhythmias and the ICD/CRTds' interventions, and to prevent mortality events in these' patients. On other hand, still a higher percentage of patients result as non responders to an ablative approach with higher acute and long term mortality rate. Therefore, in the present study in a population of HF patients (DM vs. non DM patients) affected by VA, authors will investigate the effects of CA on mortality rate at 12 months of follow up. In addition, authors would demonstrate the ameliorative effects of new hypoglycemic drugs in addition to CA in patients with DM. However, after CA the patients with DM will be randomly assigned to SGLT2 therapy vs. placebo. Indeed, study hypothesis will be that, a) DM vs. non DM patients might have higher mortality rate after CA; b) patients with DM treated by CA plus SLGT2 therapy vs. patients with DM treated by CA plus placebo might experience a lower rate of mortality at 1 year of follow-up.

DETAILED DESCRIPTION:
SLGT2 therapy is safety used in heart failure (HF) patients with depressed left ventricle ejection fraction (LVEF) and diabetes mellitus (DM). Indeed, in these patients SGLT2 therapy reduces hospital admission for heart failure and mortality rate. To date, these patients experience higher rate of ventricular arrhythmias (VA), that are a leading cause of cardiac arrest and mortality. However, as indicated by international guidelines, these patients can be treated by implantable cardioverter defibrillator (ICD) and CRTd as primary and/or secondary prevention therapy. Consequently, the effectiveness of ICD and CRTd is to treat sustained VA, and to reduce cardiac arrest events and mortality. Indeed, ICDs/CRTds' anti-tachycardia pacing and shocks can interrupt VA, and this might prevent a cardiac arrest event. This therapeutic effect can positively impact on acute and long term patients' survival. On other hand, authors showed that, continuous VA events and ICDs' interventions are causes of reduced patients' life expectancy in HF patients. This worse prognosis is particularly evidenced in failing heart patients with DM as compared to patients without DM. In this setting, the catheter ablation (CA) treatment has been used to reduce the ventricular arrhythmias and the ICDs/CRTds' interventions, and to prevent mortality events in these patients. On other hand, still a higher percentage of patients result as non responders to an ablative approach with higher acute and long term mortality rate. Among these non responders patients to an ablative approach, DM is a negative prognostic factor. Therefore, in the present study in a population of HF patients (DM vs. non DM patients) with VA authors will investigate the effects of CA on mortality rate at 12 months of follow up. In addition, authors would like to demonstrate the ameliorative effects of new hypoglycemic drugs in addition to CA in patients with DM. However, after CA the patients with DM will be randomly assigned to SGLT2 therapy vs. placebo. Indeed, study hypothesis will be that, a) DM vs. non DM might have higher mortality rate after CA; b) patients with DM treated by CA plus SLGT2 therapy vs. patients with DM treated by CA plus placebo might experience a lower rate of mortality at 1 year of follow-up. Therefore, study aim will be to demonstrate a reduction of VA, ICDs/CRTds' interventions, and mortality in patients with DM treated by CA plus SLGT2 therapy vs. patients with DM treated by CA plus placebo at 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* heart failure (HF) under optimal maximal drug therapy with NYHA functional II-III;
* HF with prior echocardiographic evidence of left ventricular systolic dysfunction (LVEF <35 % or subjective assessment of LV dysfunction that is mild or worse);
* patients under furosemide 80 mg daily or less, or equivalent loop diuretic;
* patients with stable HF symptoms for at least 3 months prior to consent;
* patients on stable therapy for HF for at least 3 months prior to consent;
* patients without hospitalization for HF for at least 3 months prior to consent;
* Ischemic and non ischemic dilated cardiomiopathy diagnosis;
* patients with internal cardioverter defibrillator (ICD);
* patients with cardioverter resynchronization therapy and defibrillator (CRTd);
* patients with diagnosis of diabetes mellitus (DM);
* patients aged >18 years and <75 years

Exclusion Criteria:

* Patients without ICD;
* patients without previous event of ventricular arrhythmia (VA);
* patients without indication to receive catheter ablation (CA) for VA;
* patients with type 1 diabetes mellitus;
* severe hepatic disease, renal disease defined as chronic kidney disease stage 3b or worse (i.e. glomerular filtration rate <45 ml/min);
* systolic blood pressure <95 mmHg at screening visit;
* screening HbA1c <6.0 %;
* patients unable to walk or to perform cardio pulmonary exercise testing or six minute walking test;
* malignancy (receiving active treatment) or other life threatening diseases;
* pregnant or lactating women;
* patients who have participated in any other clinical trial of an investigational medicinal product within the previous 30 days;
* patients who were unable to give informed consent;
* any other reason considered by a study physician to be inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
all cause deaths | 12 months
  after the intervention authors will evaluate all cause of deahs
cardiac deaths | 12 months
  after the intervention authors will evaluate the cause of cardiac deahs
ventricular arrhythmias recurrence | 12 months
  after the intervention authors will evaluate the cases of ventricular arrhythmias recurrences

SECONDARY OUTCOMES:
hospitalization for heart failure worsening | 12 months
  after the intervention authors will evaluate the causes of hospital re-admission for heart failure worsening

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: No